CLINICAL TRIAL: NCT06098820
Title: The Effect of Consumption of UV-C Enriched Foods on Biochemical Findings in Adults With Vitamin D Deficiency
Brief Title: The Effect of UV-C Enriched Foods on Vitamin D Deficiency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Okan University (Other)
Collaborators: Arçelik A.Ş. (Unknown)
Responsible Party: Principal Investigator, Aylin Seylam Küşümler, Assistant Professor, Okan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Screening
Other Study IDs: 2013
Record Dates: First submitted 2023-10-13; First posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Vitamin d Deficiency
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Intervention Model Description: Forty-eight people aged 18-65 years with serum 25(OH)vitamin D levels below 30 μg/L and who meet the study criteria will be selected for the study. Four groups, 12 per group, will be randomly selected by computer-assisted randomization.
  Group 1 (UV-C mushroom+normal bread group):
  Group 2 (UV-C mushroom + UV-C bread group) Group 3 (normal mushroom + normal bread group) Group 4 (normal mushroom + normal bread + supplement group)
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (UV-C mushroom+normal bread group) (Experimental): UV-C mushroom+normal bread group
  Interventions: Other: Vitamin D status
- Group 2 (UV-C mushroom + UV-C bread group) (Experimental): UV-C mushroom + UV-C bread group
  Interventions: Other: Vitamin D status
- Group 3 (normal mushroom + normal bread group) (Experimental): normal mushroom + normal bread group
  Interventions: Other: Vitamin D status
- Group 4 (normal mushroom+normal bread+supplemente group) (Experimental): normal mushroom + normal bread + supplement group
  Interventions: Other: Vitamin D status

INTERVENTIONS:
Other: Vitamin D status — Four different groups will be compared with each other in terms of vitamin D effect.

SUMMARY:
This study is an experimental design study in which demographic characteristics, food consumption, biochemical parameters and anthropometric measurements of individuals with low vitamin D levels before and after consuming UV-enriched foods will be examined.

DETAILED DESCRIPTION:
It was designed to be applied to individuals with low vitamin D levels working in Fatih Sultan Mehmet Training and Research Hospital who meet the research conditions.

n the first phase of the study, demographic information will be recorded by asking demographic information from the people who volunteered to participate in the study and who meet the study criteria by using a questionnaire form and 3-day food consumption record information by face-to-face interview technique; anthropometric measurements of the participants will be taken and baseline blood values will be recorded. At the beginning of the experimental study, individuals will be randomized by computer-assisted randomization into four different groups. Biochemical analyses will be analyzed every two weeks, analyses will be repeated 1 month after the study and the effects of vitamin D enrichment on biochemical parameters will be determined.

ELIGIBILITY:
Inclusion Criteria:

1. Working in the hospital
2. Being between the ages of 18 and 65
3. Not being pregnant or lactating
4. Not taking vitamin D supplements or fish oil in the last 1 month
5. Serum 25(OH)vitamin D value below 30 μg/L
6. No kidney disease, kidney stones, cortisone use, blood thinners
7. Not being in a solarium
8. Not eating fish more than once a week
9. Volunteering to participate in the research

Exclusion Criteria:

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-03-05 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Vitamin D values | Pre-intervention, through study completion, an average of every two weeks and 1 month after the completion of the intervention
  During study, Vitamin D values are evaluated.
Biochemical parameters | Pre-intervention, through study completion, an average of every two weeks and 1 month after the completion of the intervention
  Ca and parathormone are evaluated during the study.
Demographic parameters | Pre-intervention
  Demographic values (age, gender, etc.) are also investigated.
Food consumption record | Pre-intervention, through study completion, an average of every two weeks and 1 month after the completion of the intervention
  Before starting the study and after the end of study the food consumption of participants are evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- OkanU, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No